CLINICAL TRIAL: NCT07305012
Title: Feasibility and Acceptability of a New Tool for a Conscious Education and Motivation Promoting a hEalthy LIfestyle in Liver and Kidney Transplant rEcipients
Brief Title: Feasibility and Acceptability of a New Tool Promoting a Healthy Lifestyle in Liver and Kidney Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Lucia Brodosi, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: ELITE-AOUBO-IT-1; 101080645 (Other Grant/Funding Number: European Commission coordinated by Luxembourg Institute of Health Department of Precision Health)
Record Dates: First submitted 2025-11-24; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplant; Kidney Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Other): The intervention to promote a healthy lifestyle, through counseling activities combined with Digital Support Tools (Nutrida and Gamebus), will be prescribed by all partecipants
  Interventions: Behavioral: Promoting a Healthy Lifestyle through Digital Support Tools (Nutrida and Gamebus)

INTERVENTIONS:
Behavioral: Promoting a Healthy Lifestyle through Digital Support Tools (Nutrida and Gamebus) — The intervention to promote a healthy lifestyle, through counseling activities combined with Digital Support Tools (Nutrida and Gamebus), will be prescribed by all partecipants

SUMMARY:
This interventional clinical trial tests whether a doctor-delivered lifestyle counseling program, supported by two personalized digital tools, is feasible and helpful for improving healthy eating and physical activity in older adults (65 years or older) who previously received a liver or kidney transplant.

All participants first receive medical counseling on healthy diet and physical activity. After 12 weeks, they begin using two smartphone apps ("Gamebus" and "Nutrida") designed to support behavior change at home. Each participant acts as their own comparison, and results after starting the apps are compared with their own results before using them.

The main goal is to find out whether participants can safely use the apps and follow the program (for example: staying in the study, using the apps daily, completing weekly tasks). The study also looks at whether the combined approach-counseling plus digital support-can help improve eating habits, physical activity, body measurements, and routine lab values related to metabolic health.

Participants attend three study visits over 24 weeks. At each visit, they complete questionnaires, undergo body measurements and body composition tests, review their recent diet, and receive lifestyle guidance. At the end, the study will help determine whether this digital-supported lifestyle program is practical and acceptable for older transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Liver or kidney transplant received at least 6 months and no more than 25 years prior
* BMI between 21 and 29.9
* Signed informed consent
* Having a personal smartphone
* Stable immunosuppressive therapy in the past 3 months

Exclusion Criteria:

* Significant weight change (>5% of body weight) in the past 3 months
* Combined liver-kidney transplant
* Medical conditions requiring specific diets that may render adherence to the dietary recommendations of the trial unsafe (e.g., chronic kidney disease, inflammatory bowel disease, celiac disease, bariatric surgery, etc.)
* General physical conditions deemed by the investigator to contraindicate safe participation in any of the trial activities (e.g., blindness, vertebral fractures, wheelchair dependence, home oxygen therapy, etc.)
* Adherence to specific dietary regimens for ethical and/or religious reasons that are incompatible with the dietary recommendations of this trial
* Active malignant tumors currently under pharmacological treatment or awaiting surgical treatment (except cutaneous squamous cell carcinomas), or history of malignant tumors within the last 5 years, except for hepatocellular carcinoma
* Psychiatric comorbidities deemed by the investigator to potentially compromise safety and/or adherence, thereby risking biasing the results (e.g., schizophrenia, bipolar disorder, eating disorders, etc.)
* Changes in glucose-lowering or lipid-lowering therapy during the 90 days prior to the enrollment visit
* Active participation in another research or non-research program aimed at lifestyle modification
* Any clinical condition, diagnosed or under diagnostic evaluation, that the investigator considers may compromise safety and/or a priori adherence to the intervention, with a potential risk of altering the study outcomes

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to a Personalized Digital-Mediated Lifestyle Intervention in Transplant Recipients Aged ≥65 Years | Between weeks 12 and 24 from the enrollment
  Adherence will be measured between weeks 12 and 24 through the following criteria: dropout rate <5%, daily use of each app >5 minutes, >2 daily log-ins per app, and >4 weekly tasks completed in the "Gamebus" app.

SECONDARY OUTCOMES:
Effect of the Integrated Digital Intervention on Adherence to a Healthy Dietary Pattern | At weeks 12 and 24
  The effect of the intervention on dietary adherence will be evaluated through changes in Mediterranean diet adherence assessed via MEDAS score categories
Effect of the Integrated Digital Intervention on Physical Activity | At weeks 12 and 24
  The effect on physical activity will be evaluated by the number of participants with age-normative handgrip strength (in kg) values being equal to or greater than baseline.
Effect of the Integrated Intervention on Body Composition and Anthropometric Parameters | At baseline, 12 week, and 24 week.
  Variations in fat mass (%)
Effect of the Integrated Intervention on Glycolipid Metabolic Parameters | At baseline, 12 weeks, and 24 weeks.
  Changes in triglycerides (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No